CLINICAL TRIAL: NCT00196976
Title: Evaluate the Immunogenicity, Reactogenicity, Safety of 4 Different Formulations of GSK Biologicals' Conjugate Vaccine (MenACWY) vs 1 Dose of MenC-CRM197 or Mencevax™ ACWY in Children Aged 12-14 Months & 3-5 Years
Brief Title: Safety & Immunogenicity of 1 Dose of GSK134612 in Children 12-14 Months and 3-5 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103533; 103534 (Other: GSK)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-04

CONDITIONS: Infections, Meningococcal
Keywords: Safety; Meningococcal vaccine; Dose selection; Toddlers; Immunogenicity; Conjugate vaccine; Reactogenicity; Children
MeSH Terms: conditions — Meningococcal Infections | interventions — Vaccines; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Care Provider

ARMS (14):
- GSK134612A Form1 (T), Primary Group (Experimental): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, were administered one dose of formulation 1 (Form1) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533). In accordance with local immunization policy, one dose of a diphtheria, tetanus and acellular pertusis (Infanrix™ or Infanrix™ Hexa) vaccine was also administered intramuscularly into the left thigh, one month after meningococcal vaccination.
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™); Biological: Mencevax™ACWY
- GSK134612A Form2 (T), Primary Group (Experimental): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, were administered one dose of formulation 2 (Form2) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533). In accordance with local immunization policy, one dose of a diphtheria, tetanus and acellular pertusis (Infanrix™ or Infanrix™ Hexa) vaccine was also administered intramuscularly into the left thigh, one month after meningococcal vaccination.
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- GSK134612A Form3 (T), Primary Group (Experimental): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, were administered one dose of formulation 3 (Form3) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533). In accordance with local immunization policy, one dose of a diphtheria, tetanus and acellular pertusis (Infanrix™ or Infanrix™ Hexa) vaccine was also administered intramuscularly into the left thigh, one month after meningococcal vaccination.
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- GSK134612A Form4 (T), Primary Group (Experimental): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, were administered one dose of formulation 4 (Form4) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533). In accordance with local immunization policy, one dose of a diphtheria, tetanus and acellular pertusis (Infanrix™ or Infanrix™ Hexa) vaccine was also administered intramuscularly into the left thigh, one month after meningococcal vaccination.
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- Control (T), Primary Group (Active Comparator): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, were administered one dose of Pfizer's Meningitec™ conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533). In accordance with local immunization policy, one dose of a diphtheria, tetanus and acellular pertusis (Infanrix™ or Infanrix™ Hexa) vaccine was also administered intramuscularly into the left thigh, one month after meningococcal vaccination.
  Interventions: Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™); Biological: Meningitec™; Biological: Mencevax™ACWY
- GSK134612A Form1 (C), Primary Group (Experimental): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 1 (Form1) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- GSK134612A Form2 (C), Primary Group (Experimental): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 2 (Form2) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- GSK134612A Form3 (C), Primary Group (Experimental): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 3 (Form3) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- GSK134612A Form4 (C), Primary Group (Experimental): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 4 (Form4) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib); Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™)
- Control (C), Primary Group (Active Comparator): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of Mencevax™ ACWY vaccine, subcutaneously into the left upper arm, during this primary vaccination study (103533).
  Interventions: Biological: Mencevax™ACWY
- GSK134612A Form1 (T), Booster Group (Experimental): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, who 12 months after being primed with formulation 1 (Form1) of the GSK134612A conjugate vaccine, additionally received 1/5 dose of Mencevax™ ACWY vaccine subcutaneously into the left upper arm, during the booster study (103534).
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine); Biological: Mencevax™ACWY
- Control (T), Booster Group (Active Comparator): Healthy male and female toddlers (T) between, and including, 12 to 14 months of age at the time of the first vaccination, who 12 months after being primed with Pfizer's Meningitec™ conjugate vaccine, additionally received 1/5 dose of Mencevax™ ACWY vaccine subcutaneously into the left upper arm, during the booster study (103534).
  Interventions: Biological: Meningitec™; Biological: Mencevax™ACWY
- GSK134612A Form1 (C), Booster Group (Experimental): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, who 12 months after being primed with formulation 1 (Form1) of the GSK134612A conjugate vaccine, did not receive any booster vaccination.
  Interventions: Biological: Conjugated meningococcal ACWY-TT (vaccine)
- Control (C), Booster Group (Active Comparator): Healthy male and female children (C) between, and including, 3 to 5 years of age at the time of the first vaccination, who 12 months after being primed with Pfizer's Meningitec™ conjugate vaccine, did not receive any booster vaccination.
  Interventions: Biological: Meningitec™

INTERVENTIONS:
Biological: Conjugated meningococcal ACWY-TT (vaccine) — One intramuscular dose during the primary vaccination
  Arms: GSK134612A Form1 (C), Booster Group; GSK134612A Form1 (C), Primary Group; GSK134612A Form1 (T), Booster Group; GSK134612A Form1 (T), Primary Group; GSK134612A Form2 (C), Primary Group; GSK134612A Form2 (T), Primary Group; GSK134612A Form3 (C), Primary Group; GSK134612A Form3 (T), Primary Group; GSK134612A Form4 (C), Primary Group; GSK134612A Form4 (T), Primary Group
Biological: DTPa-IPV/Hib vaccine (Infanrix™-IPV/Hib) — One intramuscular dose during the primary vaccination study in subjects of 12-24 months of age, in Greece only
  Arms: Control (T), Primary Group; GSK134612A Form1 (C), Primary Group; GSK134612A Form1 (T), Primary Group; GSK134612A Form2 (C), Primary Group; GSK134612A Form2 (T), Primary Group; GSK134612A Form3 (C), Primary Group; GSK134612A Form3 (T), Primary Group; GSK134612A Form4 (C), Primary Group; GSK134612A Form4 (T), Primary Group
Biological: DTPa-HBV-IPV/Hib vaccine (Infanrix hexa™) — One intramuscular dose during the primary vaccination study in subjects of 12-24 months of age, in Austria only
  Arms: Control (T), Primary Group; GSK134612A Form1 (C), Primary Group; GSK134612A Form1 (T), Primary Group; GSK134612A Form2 (C), Primary Group; GSK134612A Form2 (T), Primary Group; GSK134612A Form3 (C), Primary Group; GSK134612A Form3 (T), Primary Group; GSK134612A Form4 (C), Primary Group; GSK134612A Form4 (T), Primary Group
Biological: Meningitec™ — One intramuscular dose during the primary vaccination study in subjects of 12-24 months of age
  Arms: Control (C), Booster Group; Control (T), Booster Group; Control (T), Primary Group
Biological: Mencevax™ACWY — One subcutaneous dose during the primary vaccination study in subjects of 3-5 years of age (Group E) and intramuscular administration of 1/5 dose during the booster vaccination study in subjects of 12-14 months of age (Groups A and E)
  Arms: Control (C), Primary Group; Control (T), Booster Group; Control (T), Primary Group; GSK134612A Form1 (T), Booster Group; GSK134612A Form1 (T), Primary Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of one dose of four different formulations of the MenACWY conjugate vaccine when given to healthy children aged 12-14 months and 3-5 years. The selection of the best formulation will be based on data obtained up to one month after the vaccine dose.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The study will enrol subjects of 12 to 14 months of age and subjects of 3 to 5 years of age. 3 formulations of GSK's MenACWY conjugate vaccine will be administered in a double-blind manner, while the 4th one will be single-blinded. Administration of the candidate vaccine or the active controls (MenC-CRM197 or Mencevax™ ACWY) will be done in an open manner. The study will be conducted in two stages: The primary vaccination phase (Study Stage 1) of the study will include all subjects; the second (booster/persistence) phase of the study (Study Stage 2) will include subjects in the active control groups and in the group which was primed with the selected MenACWY formulation.

The study will be conducted in a double-blind manner for groups receiving formulations A, B, C and in single blind manner with respect to the group receiving formulation D. The control vaccines will be administered in an open manner with respect to the investigational vaccination regimens.

Each group will have one blood sample prior to and one blood sample one month after the first vaccine dose.

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including 12 and 14 months or 3 and 5 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her parents'/guardians' knowledge. For pertussis vaccination, the children aged 12-14 months should have been vaccinated with an acellular pertussis vaccine.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the first dose of vaccine and up to one month after administration of each study vaccine dose with the exception of oral polio vaccine (OPV).
* Previous vaccination against meningococcal serogroup A, C, W-135 or Y disease.
* Administration of a H. influenzae type b, diphtheria or tetanus vaccine within 3 months before the first dose of vaccine.
* For subjects aged 12-14 months at enrolment:

  * For Austria: DTPa-HBV-IPV/Hib booster vaccination in the second year of life: these booster vaccines will be given at Visit 2.
  * For Greece: DTPa-IPV/Hib booster vaccination in the second year of life: these booster vaccines will be given at Visit 2.
* History of meningococcal serogroup A, C, W-135 or Y disease.
* Known exposure to meningococcal serogroup A, C, W-135 or Y disease within the previous year.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 461 (Actual)
Dates: Start 2005-03-24; Primary Completion 2006-03-01 (Actual); Study Completion 2006-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Austria (6):
  - GSK Investigational Site, Eferding
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Villach
  - GSK Investigational Site, Wels
- Greece (11):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Koufalia
  - GSK Investigational Site, Markopoulo Mesogaias
  - GSK Investigational Site, N. Efkarpia, Thessaloniki
  - GSK Investigational Site, Nea Makri
  - GSK Investigational Site, Rio/Patras
  - GSK Investigational Site, Thessaloniki
  - GSK Investigational Site, Tripoli

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 103533 are summarised with study 103534 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103533 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Primary Study
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Started | 39 | 41 | 41 | 40 | 40 | 54 | 50 | 52 | 52 | 52 | 0 | 0 | 0 | 0
Completed | 38 | 40 | 37 | 39 | 37 | 52 | 50 | 49 | 52 | 51 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 4 | 1 | 3 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Migrated from study area | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Booster Study
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 32 | 45 | 43
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 30 | 45 | 43
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group | Total
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 54 | 50 | 52 | 52 | 52 | 33 | 32 | 45 | 43 | 614
Age, Continuous [Mean (Standard Deviation); unit: Months] — Primary study
  Months | 12.5 (0.82) | 12.8 (0.86) | 12.8 (0.86) | 12.9 (0.83) | 12.8 (0.79) | 48.1 (7.12) | 48 (7.22) | 47.8 (7.01) | 48 (7.78) | 47.7 (7.15) | NA (NA) — This group was only included in the Booster study. | NA (NA) — This group was only included in the Booster study. | NA (NA) — This group was only included in the Booster study. | NA (NA) — This group was only included in the Booster study. | 32.59 (4.45)
Age, Continuous [Mean (Standard Deviation); unit: Months] — Booster study
  Months | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | NA (NA) — This group was only included in the Primary study. | 24.9 (1.24) | 24.9 (1.27) | 60.8 (7.23) | 60.0 (7.36) | 45.32 (18.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Primary study
  Participants
    Female | 15 | 15 | 17 | 24 | 19 | 21 | 16 | 23 | 27 | 27 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | 24 | 26 | 24 | 16 | 21 | 33 | 34 | 29 | 25 | 25 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants] — Booster study
  Participants
    Female | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | 11 | 15 | 16 | 23 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | 22 | 17 | 29 | 20 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Primary study
  Participants
    White/ Caucasian | 38 | 40 | 40 | 38 | 39 | 53 | 50 | 50 | 50 | 51 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Arabic/ north african | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    East/ south east asian | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Black | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — This group was only included in the Booster study. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Booster study
  Participants
    White/Caucasian | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | 32 | 31 | 44 | 43 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Arabic/north African | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | NA — This group was only included in the Primary study. | 1 | 1 | 1 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Immune Response to Different Meningococcal Serogroups
Description: A responder to serum bactericidal assay meningococcal serogroups A, C, W and Y, using rabbit complement (rSBA-MenA, rSBA-MenC, rSBA-MenW-135, rSBA-MenY) was defined as follows: -for initially seronegative subjects (antibody titers < 1:8 for rSBA-Men), a subject achieving a post-vaccination rSBA-Men antibody titer of ≥ 1:32; - for initially seropositive subjects (antibody titers ≥ 1:8 for rSBA-Men), a subject having a ≥ 4-fold increase in rSBA-Men antibody titer from pre to post vaccination.
Time Frame: One month after the first vaccine dose (Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 36 | 29 | 35 | 33 | 50 | 48 | 46 | 50 | 43
Participants
  rSBA-MenA: number analyzed (Participants) | 33 | 34 | 26 | 31 | 31 | 45 | 45 | 44 | 50 | 40
  rSBA-MenA | 30 | 32 | 26 | 27 | 6 | 41 | 38 | 41 | 42 | 36
  rSBA-MenC: number analyzed (Participants) | 32 | 34 | 29 | 34 | 32 | 50 | 48 | 46 | 49 | 42
  rSBA-MenC | 30 | 32 | 26 | 33 | 30 | 45 | 44 | 44 | 46 | 34
  rSBA-MenW-135: number analyzed (Participants) | 35 | 36 | 28 | 35 | 33 | 47 | 47 | 46 | 48 | 43
  rSBA-MenW-135 | 34 | 36 | 27 | 35 | 3 | 46 | 44 | 46 | 48 | 36
  rSBA-MenY: number analyzed (Participants) | 36 | 35 | 29 | 34 | 33 | 48 | 48 | 46 | 50 | 43
  rSBA-MenY | 33 | 34 | 26 | 34 | 3 | 46 | 47 | 45 | 47 | 34

2. Secondary Outcome: Number of Seroprotected Subjects Against Different Meningococcal Serogroups
Description: A seroprotected subject against meningococcal serogroups rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY assessed, was defined as having antibody titers greater than or equal to (≥) 1:8.
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 30 | 35 | 35 | 51 | 48 | 48 | 50 | 44
Participants
  rSBA-MenA, Month 0: number analyzed (Participants) | 33 | 34 | 27 | 32 | 34 | 46 | 46 | 44 | 50 | 41
  rSBA-MenA, Month 0 | 23 | 22 | 19 | 21 | 20 | 41 | 42 | 40 | 47 | 39
  rSBA-MenA, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 34 | 32 | 50 | 47 | 48 | 50 | 43
  rSBA-MenA, Month 1 | 36 | 38 | 30 | 34 | 23 | 50 | 47 | 48 | 50 | 43
  rSBA-MenC, Month 0: number analyzed (Participants) | 32 | 34 | 30 | 34 | 32 | 50 | 48 | 47 | 49 | 42
  rSBA-MenC, Month 0 | 5 | 2 | 2 | 5 | 3 | 16 | 8 | 17 | 12 | 14
  rSBA-MenC, Month 1: number analyzed (Participants) | 36 | 38 | 29 | 35 | 35 | 51 | 48 | 47 | 50 | 44
  rSBA-MenC, Month 1 | 36 | 38 | 28 | 35 | 34 | 50 | 47 | 47 | 49 | 43
  rSBA-MenW-135, Month 0: number analyzed (Participants) | 35 | 36 | 29 | 35 | 34 | 47 | 47 | 46 | 48 | 43
  rSBA-MenW-135, Month 0 | 17 | 19 | 12 | 13 | 15 | 34 | 24 | 25 | 36 | 27
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenW-135, Month 1 | 35 | 38 | 30 | 35 | 15 | 50 | 48 | 48 | 50 | 44
  rSBA-MenY, Month 0: number analyzed (Participants) | 36 | 35 | 30 | 34 | 34 | 48 | 48 | 46 | 50 | 43
  rSBA-MenY, Month 0 | 23 | 17 | 16 | 19 | 22 | 37 | 42 | 39 | 42 | 36
  rSBA-MenY, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenY, Month 1 | 35 | 38 | 29 | 35 | 25 | 51 | 48 | 48 | 50 | 44

3. Secondary Outcome: Number of Seropositive Subjects for Different Anti-meningococcal Serogroups
Description: A seropositive subject for meningococcal serogroups rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-Y assessed, was defined as having antibody titers greater than or equal to (≥) 1:128.
Time Frame: Prior to (Month 0) and one month after (Month 1) after the first vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 30 | 35 | 35 | 51 | 48 | 48 | 50 | 44
Participants
  rSBA-MenA, Month 0: number analyzed (Participants) | 33 | 34 | 27 | 32 | 34 | 46 | 46 | 44 | 50 | 41
  rSBA-MenA, Month 0 | 19 | 19 | 13 | 19 | 17 | 41 | 39 | 40 | 46 | 37
  rSBA-MenA, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 34 | 32 | 50 | 47 | 48 | 50 | 43
  rSBA-MenA, Month 1 | 36 | 38 | 29 | 34 | 20 | 49 | 47 | 48 | 50 | 43
  rSBA-MenC, Month 0: number analyzed (Participants) | 32 | 34 | 30 | 34 | 32 | 50 | 48 | 47 | 49 | 42
  rSBA-MenC, Month 0 | 3 | 0 | 0 | 3 | 1 | 9 | 4 | 5 | 7 | 5
  rSBA-MenC, Month 1: number analyzed (Participants) | 36 | 38 | 29 | 35 | 35 | 51 | 48 | 47 | 50 | 44
  rSBA-MenC, Month 1 | 35 | 34 | 26 | 31 | 27 | 49 | 46 | 45 | 48 | 39
  rSBA-MenW-135, Month 0: number analyzed (Participants) | 35 | 36 | 29 | 35 | 34 | 47 | 47 | 46 | 48 | 43
  rSBA-MenW-135, Month 0 | 8 | 9 | 4 | 4 | 8 | 19 | 11 | 9 | 15 | 12
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenW-135, Month 1 | 35 | 38 | 29 | 35 | 9 | 50 | 48 | 48 | 49 | 42
  rSBA-MenY, Month 0: number analyzed (Participants) | 36 | 35 | 30 | 34 | 34 | 48 | 48 | 46 | 50 | 43
  rSBA-MenY, Month 0 | 17 | 11 | 9 | 12 | 17 | 29 | 37 | 32 | 33 | 30
  rSBA-MenY, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenY, Month 1 | 35 | 37 | 29 | 34 | 18 | 51 | 48 | 48 | 50 | 43

4. Secondary Outcome: Antibody Titers Against Different Meningococcal Serogroups
Description: Antibody titers against meningococcal serogroups A, C, W-135 and Y (MenA, MenC, MenW-135 and MenY) have been assessed, using rabbit complement and expressed as geometric mean titers (GMTs).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 30 | 35 | 35 | 51 | 48 | 48 | 50 | 44
Titers
  rSBA-MenA, Month 0: number analyzed (Participants) | 33 | 34 | 27 | 32 | 34 | 46 | 46 | 44 | 50 | 41
  rSBA-MenA, Month 0 | 84.2 [39.3 to 180.1] | 77.3 [32.9 to 181.6] | 68.4 [30.1 to 155.3] | 76 [33.8 to 170.8] | 69.1 [28.1 to 169.9] | 359.7 [212 to 610.4] | 367.2 [222.1 to 607] | 375.9 [227.4 to 621.2] | 465.2 [307.2 to 704.4] | 427.4 [280.3 to 651.7]
  rSBA-MenA, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 34 | 32 | 50 | 47 | 48 | 50 | 43
  rSBA-MenA, Month 1 | 6648 [4787.3 to 9231.9] | 5406.8 [3961.5 to 7379.4] | 6225.2 [3510.2 to 11040.2] | 3928.6 [2851.5 to 5412.4] | 125.9 [53.1 to 298.3] | 7469.5 [5468.8 to 10202.1] | 7569.7 [6044 to 9480.6] | 13668.3 [11274.3 to 16570.6] | 4878 [4002.5 to 5944.9] | 4556.8 [3598 to 5771.1]
  rSBA-MenC, Month 0: number analyzed (Participants) | 32 | 34 | 30 | 34 | 32 | 50 | 48 | 47 | 49 | 42
  rSBA-MenC, Month 0 | 6.9 [4.1 to 11.5] | 4.5 [3.8 to 5.2] | 4.6 [3.8 to 5.7] | 6.6 [4.2 to 10.2] | 5.3 [3.8 to 7.3] | 12.5 [7.6 to 20.5] | 7.4 [4.7 to 11.6] | 11.8 [7.5 to 18.5] | 8.9 [5.7 to 14.1] | 11.9 [7 to 20.2]
  rSBA-MenC, Month 1: number analyzed (Participants) | 36 | 38 | 29 | 35 | 35 | 51 | 48 | 47 | 50 | 44
  rSBA-MenC, Month 1 | 656.4 [483 to 892] | 495.7 [334.6 to 734.4] | 477.2 [245.1 to 929.4] | 464.3 [324.4 to 664.5] | 404.5 [222.5 to 735.4] | 967.6 [672 to 1393.3] | 1115 [746.4 to 1665.7] | 1738.8 [1159.7 to 2607] | 1197.6 [765 to 1874.7] | 378.3 [257.2 to 556.5]
  rSBA-MenW-135, Month 0: number analyzed (Participants) | 35 | 36 | 29 | 35 | 34 | 47 | 47 | 46 | 48 | 43
  rSBA-MenW-135, Month 0 | 19.8 [10.7 to 36.9] | 21.1 [11.5 to 38.6] | 14.5 [7.7 to 27.3] | 12.1 [7.1 to 20.6] | 18 [9.7 to 33.6] | 45.8 [27.9 to 75.2] | 22.3 [12.7 to 39] | 23.7 [14.2 to 39.7] | 44.6 [28.1 to 71] | 31.5 [18 to 55]
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenW-135, Month 1 | 2781.4 [1647 to 4697.2] | 3447.5 [2484.8 to 4783.3] | 2545 [1522.2 to 4254.9] | 3260.8 [2342.1 to 4539.8] | 21.7 [10.5 to 44.9] | 4317.4 [3114.8 to 5984.3] | 3856.5 [3153.4 to 4716.4] | 5262.1 [4417.8 to 6267.7] | 4556.1 [3576.6 to 5803.7] | 912.7 [659.1 to 1264.1]
  rSBA-MenY, Month 0: number analyzed (Participants) | 36 | 35 | 30 | 34 | 34 | 48 | 48 | 46 | 50 | 43
  rSBA-MenY, Month 0 | 57.7 [27.5 to 121.3] | 24.4 [12 to 49.7] | 32.4 [14.3 to 73] | 32.9 [15.9 to 68.3] | 52.8 [25.5 to 109.5] | 98.7 [54.9 to 177.5] | 181.9 [112.1 to 295.3] | 146.8 [86.2 to 250.1] | 140.6 [82.8 to 238.9] | 123.6 [73.3 to 208.6]
  rSBA-MenY, Month 1: number analyzed (Participants) | 36 | 38 | 30 | 35 | 34 | 51 | 48 | 48 | 50 | 44
  rSBA-MenY, Month 1 | 2599.9 [1531.8 to 4412.7] | 2150.9 [1486.2 to 3112.9] | 1920.9 [1014.2 to 3638.2] | 3544.7 [2480.2 to 5065.9] | 75.6 [38.1 to 150.1] | 5249.1 [4107.9 to 6707.4] | 5150.5 [4149.8 to 6392.6] | 5896.3 [4686.4 to 7418.5] | 7548.4 [6116.1 to 9316.2] | 1527.3 [1110.8 to 2099.9]

5. Secondary Outcome: Number of Seropositive Subjects for Different Anti-meningococcal Polysaccharides
Description: A seropositive subject for meningococcal polysaccharide A (PSA), C (PSC), W-135 (PSW-135) and Y (PSY) assessed, was defined as having antibody (anti-PSA, anti-PSC, anti-PSW-135 and anti-PSY) concentrations greater than or equal to (≥) the cut-off value of 0.3 micrograms per milliliter (μg/mL). Antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 31 | 35 | 34 | 51 | 47 | 48 | 50 | 44
Participants
  Anti-PSA, Month 0: number analyzed (Participants) | 33 | 32 | 30 | 27 | 31 | 51 | 46 | 47 | 49 | 43
  Anti-PSA, Month 0 | 1 | 2 | 0 | 1 | 0 | 10 | 4 | 6 | 9 | 10
  Anti-PSA, Month 1: number analyzed (Participants) | 36 | 36 | 31 | 34 | 30 | 48 | 46 | 48 | 49 | 44
  Anti-PSA, Month 1 | 35 | 36 | 30 | 34 | 2 | 48 | 45 | 48 | 48 | 44
  Anti-PSC, Month 0: number analyzed (Participants) | 32 | 33 | 30 | 30 | 29 | 51 | 46 | 47 | 50 | 43
  Anti-PSC, Month 0 | 1 | 1 | 0 | 1 | 1 | 3 | 4 | 1 | 1 | 2
  Anti-PSC, Month 1: number analyzed (Participants) | 34 | 38 | 31 | 35 | 34 | 49 | 46 | 48 | 49 | 44
  Anti-PSC, Month 1 | 33 | 38 | 30 | 35 | 34 | 49 | 45 | 48 | 48 | 44
  Anti-PSW-135, Month 0: number analyzed (Participants) | 34 | 35 | 30 | 33 | 33 | 51 | 47 | 48 | 50 | 44
  Anti-PSW-135, Month 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4 | 2 | 0 | 1
  Anti-PSW-135, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 35 | 34 | 50 | 46 | 48 | 49 | 44
  Anti-PSW-135, Month 1 | 34 | 36 | 30 | 35 | 0 | 48 | 45 | 48 | 48 | 44
  Anti-PSY, Month 0: number analyzed (Participants) | 34 | 36 | 30 | 32 | 34 | 51 | 47 | 48 | 50 | 44
  Anti-PSY, Month 0 | 2 | 0 | 2 | 1 | 1 | 2 | 4 | 2 | 1 | 1
  Anti-PSY, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 34 | 32 | 50 | 46 | 46 | 49 | 44
  Anti-PSY, Month 1 | 34 | 37 | 30 | 34 | 2 | 49 | 45 | 46 | 48 | 44

6. Secondary Outcome: Number of Seroprotected Subjects Against Different Meningococcal Polysaccharides
Description: A seroprotected subject for meningococcal polysaccharide A (PSA), C (PSC), W-135 (PSW-135) and Y (PSY) assessed, was defined as having antibody (anti-PSA, anti-PSC, anti-PSW-135 and anti-PSY) concentrations greater than or equal to (≥) the value of 2.0 micrograms per milliliter (μg/mL). Antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 31 | 35 | 34 | 51 | 47 | 48 | 50 | 44
Participants
  Anti-PSA, Month 0: number analyzed (Participants) | 33 | 32 | 30 | 27 | 31 | 51 | 46 | 47 | 49 | 43
  Anti-PSA, Month 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 5
  Anti-PSA, Month 1: number analyzed (Participants) | 36 | 36 | 31 | 34 | 30 | 48 | 46 | 48 | 49 | 44
  Anti-PSA, Month 1 | 35 | 35 | 30 | 25 | 0 | 48 | 44 | 47 | 34 | 40
  Anti-PSC, Month 0: number analyzed (Participants) | 32 | 33 | 30 | 30 | 29 | 51 | 46 | 47 | 50 | 43
  Anti-PSC, Month 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2
  Anti-PSC, Month 1: number analyzed (Participants) | 34 | 38 | 31 | 35 | 34 | 49 | 46 | 48 | 49 | 44
  Anti-PSC, Month 1 | 33 | 37 | 29 | 34 | 33 | 44 | 45 | 45 | 47 | 44
  Anti-PSW-135, Month 0: number analyzed (Participants) | 34 | 35 | 30 | 33 | 33 | 51 | 47 | 48 | 50 | 44
  Anti-PSW-135, Month 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Anti-PSW-135, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 35 | 34 | 50 | 46 | 48 | 49 | 44
  Anti-PSW-135, Month 1 | 33 | 27 | 23 | 32 | 0 | 41 | 31 | 41 | 39 | 39
  Anti-PSY, Month 0: number analyzed (Participants) | 34 | 36 | 30 | 32 | 34 | 51 | 47 | 48 | 50 | 44
  Anti-PSY, Month 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
  Anti-PSY, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 34 | 32 | 50 | 46 | 46 | 49 | 44
  Anti-PSY, Month 1 | 34 | 34 | 27 | 33 | 0 | 46 | 40 | 39 | 47 | 42

7. Secondary Outcome: Antibody Concentrations Against Different Meningococcal Polysaccharides
Description: The meningococcal polysaccharides assessed included polysaccharide A (anti-PSA), polysaccharide B (anti-PSB), polysaccharide W-135 (anti-PSW-135) and polysaccharide Y (anti-PSY). Antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 38 | 31 | 35 | 34 | 51 | 47 | 48 | 50 | 44
μg/mL
  Anti-PSA, Month 0: number analyzed (Participants) | 33 | 32 | 30 | 27 | 31 | 51 | 46 | 47 | 49 | 43
  Anti-PSA, Month 0 | 0.16 [0.14 to 0.18] | 0.16 [0.14 to 0.19] | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.15] | 0.2 [0.17 to 0.25] | 0.17 [0.15 to 0.2] | 0.17 [0.15 to 0.19] | 0.21 [0.17 to 0.26] | 0.25 [0.18 to 0.35]
  Anti-PSA, Month 1: number analyzed (Participants) | 36 | 36 | 31 | 34 | 30 | 48 | 46 | 48 | 49 | 44
  Anti-PSA, Month 1 | 30.65 [19.83 to 47.38] | 22.09 [16.35 to 29.84] | 34.68 [21.7 to 55.42] | 4.03 [2.72 to 5.98] | 0.17 [0.14 to 0.2] | 20.01 [14.53 to 27.56] | 12.62 [8.74 to 18.22] | 24.69 [19.14 to 31.85] | 3.63 [2.62 to 5.04] | 13.79 [9.04 to 21.02]
  Anti-PSC, Month 0: number analyzed (Participants) | 32 | 33 | 30 | 30 | 29 | 51 | 46 | 47 | 50 | 43
  Anti-PSC, Month 0 | 0.16 [0.14 to 0.17] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.17] | 0.18 [0.15 to 0.22] | 0.18 [0.15 to 0.23] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.16] | 0.18 [0.14 to 0.22]
  Anti-PSC, Month 1: number analyzed (Participants) | 34 | 38 | 31 | 35 | 34 | 49 | 46 | 48 | 49 | 44
  Anti-PSC, Month 1 | 10.67 [7.47 to 15.23] | 11.23 [8.75 to 14.4] | 12.91 [8.83 to 18.88] | 10.74 [8.43 to 13.68] | 11.99 [9.26 to 15.53] | 6.33 [4.81 to 8.34] | 7.76 [5.76 to 10.44] | 7.71 [6.05 to 9.83] | 7.78 [5.83 to 10.38] | 14.44 [11.32 to 18.42]
  Anti-PSW-135, Month 0: number analyzed (Participants) | 34 | 35 | 30 | 33 | 33 | 51 | 47 | 48 | 50 | 44
  Anti-PSW-135, Month 0 | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.17] | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.16] | 0.17 [0.15 to 0.2] | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.15] | 0.16 [0.14 to 0.17]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 35 | 34 | 50 | 46 | 48 | 49 | 44
  Anti-PSW-135, Month 1 | 7.52 [4.97 to 11.36] | 3.12 [2.3 to 4.22] | 3.62 [2.31 to 5.68] | 7.09 [5.19 to 9.7] | 0.15 [0.15 to 0.15] | 4.76 [3.4 to 6.66] | 3.2 [2.33 to 4.39] | 3.85 [2.85 to 5.21] | 4.99 [3.7 to 6.73] | 7.93 [5.39 to 11.66]
  Anti-PSY, Month 0: number analyzed (Participants) | 34 | 36 | 30 | 32 | 34 | 51 | 47 | 48 | 50 | 44
  Anti-PSY, Month 0 | 0.16 [0.14 to 0.18] | 0.15 [0.15 to 0.15] | 0.16 [0.15 to 0.17] | 0.16 [0.14 to 0.2] | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.18] | 0.19 [0.15 to 0.24] | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.16] | 0.15 [0.15 to 0.16]
  Anti-PSY, Month 1: number analyzed (Participants) | 35 | 37 | 31 | 34 | 32 | 50 | 46 | 46 | 49 | 44
  Anti-PSY, Month 1 | 10.86 [7.41 to 15.92] | 6.71 [5.12 to 8.8] | 6.01 [4 to 9.03] | 13.38 [9.48 to 18.89] | 0.16 [0.15 to 0.17] | 9.41 [6.66 to 13.31] | 6.59 [4.7 to 9.25] | 5.75 [4.23 to 7.81] | 11.7 [8.39 to 16.32] | 18.96 [13.68 to 26.29]

8. Secondary Outcome: Number of Seropositive Subjects for Anti-tetanus (Anti-T)
Description: A seropositive subject for anti-tetanus was defined as having antibody concentrations greater than or equal to (≥) the cut-off value of 0.1 international units per milliliter (IU/mL). Antibody titers were determined by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 37 | 30 | 35 | 35 | 51 | 48 | 48 | 50 | 44
Participants
  Anti-T, Month 0: number analyzed (Participants) | 35 | 36 | 30 | 33 | 34 | 51 | 48 | 48 | 50 | 44
  Anti-T, Month 0 | 34 | 36 | 30 | 32 | 33 | 49 | 47 | 46 | 48 | 43
  Anti-T, Month 1: number analyzed (Participants) | 36 | 37 | 30 | 35 | 35 | 49 | 47 | 48 | 50 | 44
  Anti-T, Month 1 | 36 | 37 | 30 | 35 | 34 | 48 | 47 | 48 | 50 | 43

9. Secondary Outcome: Antibody Concentrations Against Tetanus (Anti-T)
Description: Antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) method, presented as geometric mean concentrations (GMCs) and expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (Month 0) and one month after (Month 1) the first vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Groups:
- GSK134612A Form1 (C), Primary Group: Healthy male and female childrens (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 1 (Form1) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
- GSK134612A Form2 (C), Primary Group: Healthy male and female childrens (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 2 (Form2) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
- GSK134612A Form3 (C), Primary Group: Healthy male and female childrens (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 3 (Form3) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
- GSK134612A Form4 (C), Primary Group: Healthy male and female childrens (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of formulation 4 (Form4) of the GSK134612A conjugate vaccine, intramuscularly into the left arm's deltoid region, during this primary vaccination study (103533).
- Control (C), Primary Group: Healthy male and female childrens (C) between, and including, 3 to 5 years of age at the time of the first vaccination, were administered one dose of Mencevax™ ACWY vaccine, subcutaneously into the left upper arm, during this primary vaccination study (103533).
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 36 | 37 | 30 | 35 | 35 | 51 | 48 | 48 | 50 | 44
IU/mL
  Anti-T, Month 0: number analyzed (Participants) | 35 | 36 | 30 | 33 | 34 | 51 | 48 | 48 | 50 | 44
  Anti-T, Month 0 | 1.007 [0.671 to 1.51] | 1.159 [0.814 to 1.65] | 1.203 [0.871 to 1.662] | 1.293 [0.826 to 2.023] | 0.792 [0.578 to 1.084] | 1.426 [0.94 to 2.164] | 1.312 [0.935 to 1.841] | 1.232 [0.849 to 1.788] | 1.18 [0.823 to 1.694] | 1.083 [0.742 to 1.58]
  Anti-T, Month 1: number analyzed (Participants) | 36 | 37 | 30 | 35 | 35 | 49 | 47 | 48 | 50 | 44
  Anti-T, Month 1 | 7.559 [5.04 to 11.335] | 5.353 [3.832 to 7.477] | 8.094 [4.855 to 13.492] | 7.675 [4.783 to 12.315] | 0.696 [0.52 to 0.932] | 17.284 [11.812 to 25.292] | 15.823 [11.728 to 21.348] | 19.369 [13.226 to 28.363] | 15.957 [11.767 to 21.639] | 1.231 [0.833 to 1.82]

10. Secondary Outcome: Number of Toddlers With Any Solicited Local Symptoms
Description: The toddlers subgroup received 2 primary vaccine doses, as follows: first dose of a meningococcal vaccine and second dose of a diphtheria, tetanus and acellular pertusis-containing vaccine. Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after each primary vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who had filled in the symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 39
Participants
  Pain, Dose 1 | 4 | 8 | 3 | 6 | 4
  Redness, Dose 1 | 9 | 12 | 10 | 9 | 11
  Swelling, Dose 1 | 1 | 6 | 7 | 6 | 4
  Pain, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Pain, Dose 2 | 3 | 10 | 6 | 7 | 6
  Redness, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Redness, Dose 2 | 7 | 13 | 9 | 8 | 7
  Swelling, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Swelling, Dose 2 | 3 | 7 | 9 | 7 | 3

11. Secondary Outcome: Number of Children With Any Solicited Local Symptoms
Description: The children subgroup received one dose of the meningococcal vaccine. Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after each primary vaccine dose
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 52 | 50 | 50 | 52 | 51
Participants
  Pain | 10 | 11 | 9 | 11 | 13
  Redness | 9 | 11 | 10 | 9 | 7
  Swelling | 7 | 9 | 8 | 10 | 4

12. Secondary Outcome: Number of Toddlers With Any Solicited General Symptoms
Description: The toddlers subgroup received 2 primary vaccine doses, as follows: first dose of a meningococcal vaccine and second dose of a diphtheria, tetanus and acellular pertusis-containing vaccine. Assessed solicited general symptoms included drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = incidence of a particular symptom regardless of intensity or relationship to vaccination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after each primary vaccine dose
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 39
Participants
  Drowsiness, Dose 1 | 1 | 5 | 4 | 4 | 5
  Fever (Axillary), Dose 1 | 5 | 8 | 8 | 3 | 5
  Irritability, Dose 1 | 4 | 9 | 6 | 5 | 5
  Loss of appetite, Dose 1 | 1 | 6 | 5 | 3 | 6
  Drowsiness, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Drowsiness, Dose 2 | 2 | 2 | 3 | 7 | 3
  Fever (Axillary), Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Fever (Axillary), Dose 2 | 4 | 5 | 5 | 5 | 8
  Irritability, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Irritability, Dose 2 | 6 | 7 | 3 | 9 | 5
  Loss of appetite, Dose 2: number analyzed (Participants) | 38 | 39 | 37 | 39 | 37
  Loss of appetite, Dose 2 | 4 | 3 | 2 | 6 | 2

13. Secondary Outcome: Number of Children With Any Solicited General Symptoms
Description: The children subgroup received one primary meningococcal vaccine dose. Assessed solicited general symptoms included drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = incidence of a particular symptom regardless of intensity or relationship to vaccination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period after each primary vaccine dose
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 52 | 50 | 50 | 52 | 51
Participants
  Drowsiness | 4 | 2 | 0 | 5 | 4
  Fever (Axillary) | 4 | 4 | 3 | 3 | 3
  Irritability | 2 | 4 | 2 | 4 | 7
  Loss of appetite | 2 | 3 | 2 | 6 | 3

14. Secondary Outcome: Number of Seroprotected Subjects Against Different Meningococcal Serogroups
Description: as for outcome 2
Time Frame: At one month (M1) and 12 months (M12) post-primary vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) Cohort for antibody persistence, which included subjects primed with the selected GSK134612A formulation or the control vaccine in both age strata, for whom assay results were available for antibodies against at least one study vaccine antigen component for the Month 12 blood sampling.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 44 | 37
Participants
  rSBA-MenA, Month 1: number analyzed (Participants) | 31 | 27 | 43 | 36
  rSBA-MenA, Month 1 | 31 | 18 | 43 | 36
  rSBA-MenC, Month 1 | 31 | 29 | 43 | 36
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenW-135, Month 1 | 30 | 11 | 43 | 37
  rSBA-MenY, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenY, Month 1 | 30 | 20 | 44 | 37
  rSBA-MenA, Month 12: number analyzed (Participants) | 23 | 25 | 39 | 33
  rSBA-MenA, Month 12 | 23 | 20 | 39 | 33
  rSBA-MenC, Month 12: number analyzed (Participants) | 31 | 29 | 41 | 32
  rSBA-MenC, Month 12 | 29 | 25 | 40 | 22
  rSBA-MenW-135, Month 12: number analyzed (Participants) | 31 | 27 | 41 | 35
  rSBA-MenW-135, Month 12 | 30 | 11 | 41 | 31
  rSBA-MenY, Month 12: number analyzed (Participants) | 31 | 29 | 41 | 37
  rSBA-MenY, Month 12 | 31 | 23 | 41 | 36

15. Secondary Outcome: Number of Seropositive Subjects for Different Anti-meningococcal Serogroups
Description: as for outcome 3
Time Frame: At one month (M1) and 12 months (M12) post-primary vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 44 | 37
Participants
  rSBA-MenA, Month 1: number analyzed (Participants) | 31 | 27 | 43 | 36
  rSBA-MenA, Month 1 | 31 | 14 | 42 | 36
  rSBA-MenC, Month 1 | 31 | 23 | 42 | 34
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenW-135, Month 1 | 30 | 6 | 43 | 35
  rSBA-MenY, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenY, Month 1 | 30 | 13 | 44 | 36
  rSBA-MenA, Month 12: number analyzed (Participants) | 23 | 25 | 39 | 33
  rSBA-MenA, Month 12 | 23 | 19 | 39 | 32
  rSBA-MenC, Month 12: number analyzed (Participants) | 31 | 29 | 41 | 32
  rSBA-MenC, Month 12 | 13 | 15 | 27 | 10
  rSBA-MenW-135, Month 12: number analyzed (Participants) | 31 | 27 | 41 | 35
  rSBA-MenW-135, Month 12 | 27 | 6 | 41 | 27
  rSBA-MenY, Month 12 | 30 | 17 | 40 | 32

16. Secondary Outcome: Antibody Titers Against Different Meningococcal Serogroups
Description: as for outcome 4
Time Frame: At one month (M1) and 12 months (M12) post-primary vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 44 | 37
Titers
  rSBA-MenA, Month 1: number analyzed (Participants) | 31 | 27 | 43 | 36
  rSBA-MenA, Month 1 | 6577.8 [4606.7 to 9392.4] | 84.9 [32.4 to 222.8] | 6565.3 [4616.3 to 9337.2] | 4649.5 [3572.8 to 6050.8]
  rSBA-MenC, Month 1 | 660.4 [484.4 to 900.3] | 440.2 [227.1 to 853.1] | 893.6 [600.3 to 1330.3] | 416.2 [270.5 to 640.5]
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenW-135, Month 1 | 2523.5 [1433.1 to 4443.7] | 17.2 [7.9 to 37.8] | 3893.6 [2671.2 to 5675.6] | 1004.4 [690.4 to 1461.2]
  rSBA-MenY, Month 1: number analyzed (Participants) | 31 | 29 | 44 | 37
  rSBA-MenY, Month 1 | 2483.9 [1363.8 to 4524.1] | 57.7 [27.1 to 123.2] | 4808.5 [3653 to 6329.6] | 1641.1 [1131.2 to 2380.9]
  rSBA-MenA, Month 12: number analyzed (Participants) | 23 | 25 | 39 | 33
  rSBA-MenA, Month 12 | 2369.1 [1642 to 3418.2] | 179.3 [76.1 to 422.9] | 2356.7 [1786.7 to 3108.4] | 1134.3 [767.8 to 1675.5]
  rSBA-MenC, Month 12: number analyzed (Participants) | 31 | 29 | 41 | 32
  rSBA-MenC, Month 12 | 110.2 [60.6 to 200.7] | 122 [59 to 252.2] | 172.5 [117.7 to 252.9] | 41.7 [22 to 79.2]
  rSBA-MenW-135, Month 12: number analyzed (Participants) | 31 | 27 | 41 | 35
  rSBA-MenW-135, Month 12 | 541.8 [305.5 to 961] | 18.9 [8.4 to 42.9] | 1322.2 [978.3 to 1786.8] | 181.7 [104.6 to 315.8]
  rSBA-MenY, Month 12: number analyzed (Participants) | 31 | 29 | 41 | 37
  rSBA-MenY, Month 12 | 740.3 [493.4 to 1110.9] | 110.6 [51.6 to 237.1] | 1400.8 [1008.8 to 1945.1] | 347.2 [228.2 to 528.5]

17. Secondary Outcome: Number of Seropositive Subjects for Different Anti-meningococcal Polysaccharides
Description: as for outcome 5
Time Frame: At one month (M1) and 12 months (M12) post-primary vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 43 | 37
Participants
  Anti-PSA, Month 1: number analyzed (Participants) | 31 | 25 | 41 | 37
  Anti-PSA, Month 1 | 30 | 1 | 41 | 37
  Anti-PSC, Month 1: number analyzed (Participants) | 29 | 30 | 42 | 37
  Anti-PSC, Month 1 | 28 | 30 | 42 | 37
  Anti-PSW-135, Month 1: number analyzed (Participants) | 30 | 29 | 43 | 37
  Anti-PSW-135, Month 1 | 29 | 0 | 41 | 37
  Anti-PSY, Month 1: number analyzed (Participants) | 30 | 27 | 43 | 37
  Anti-PSY, Month 1 | 29 | 2 | 42 | 37
  Anti-PSA, Month 12: number analyzed (Participants) | 27 | 22 | 38 | 36
  Anti-PSA, Month 12 | 22 | 2 | 34 | 34
  Anti-PSC, Month 12: number analyzed (Participants) | 27 | 27 | 39 | 37
  Anti-PSC, Month 12 | 13 | 18 | 18 | 36
  Anti-PSW-135, Month 12: number analyzed (Participants) | 25 | 21 | 37 | 34
  Anti-PSW-135, Month 12 | 25 | 3 | 34 | 32
  Anti-PSY, Month 12: number analyzed (Participants) | 26 | 21 | 37 | 35
  Anti-PSY, Month 12 | 26 | 3 | 34 | 35

18. Secondary Outcome: Number of Seroprotected Subjects Against Different Meningococcal Polysaccharides
Description: as for outcome 6
Time Frame: At one month (M1) and 12 months (M12) post primary vaccination
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 43 | 37
Participants
  Anti-PSA, Month 1: number analyzed (Participants) | 31 | 25 | 41 | 37
  Anti-PSA, Month 1 | 30 | 0 | 41 | 33
  Anti-PSC, Month 1: number analyzed (Participants) | 29 | 30 | 42 | 37
  Anti-PSC, Month 1 | 28 | 29 | 37 | 37
  Anti-PSW-135, Month 1: number analyzed (Participants) | 30 | 29 | 43 | 37
  Anti-PSW-135, Month 1 | 28 | 0 | 34 | 32
  Anti-PSY, Month 1: number analyzed (Participants) | 30 | 27 | 43 | 37
  Anti-PSY, Month 1 | 29 | 0 | 39 | 35
  Anti-PSA, Month 12: number analyzed (Participants) | 27 | 22 | 38 | 36
  Anti-PSA, Month 12 | 10 | 0 | 12 | 22
  Anti-PSC, Month 12: number analyzed (Participants) | 27 | 27 | 39 | 37
  Anti-PSC, Month 12 | 2 | 4 | 0 | 24
  Anti-PSW-135, Month 12: number analyzed (Participants) | 25 | 21 | 37 | 34
  Anti-PSW-135, Month 12 | 6 | 2 | 10 | 23
  Anti-PSY, Month 12: number analyzed (Participants) | 26 | 21 | 37 | 35
  Anti-PSY, Month 12 | 15 | 1 | 19 | 30

19. Secondary Outcome: Antibody Concentrations Against Different Meningococcal Polysaccharides
Description: as for outcome 7
Time Frame: At one month (M1) and 12 months (M12) post-primary vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 31 | 30 | 43 | 37
µg/mL
  Anti-PSA, Month 1: number analyzed (Participants) | 31 | 25 | 41 | 37
  Anti-PSA, Month 1 | 32.72 [20.12 to 53.22] | 0.17 [0.14 to 0.2] | 18.29 [12.86 to 26.01] | 13 [8.19 to 20.63]
  Anti-PSC, Month 1: number analyzed (Participants) | 29 | 30 | 42 | 37
  Anti-PSC, Month 1 | 11.25 [7.48 to 16.93] | 12.43 [9.28 to 16.65] | 5.64 [4.21 to 7.57] | 14.5 [11.01 to 19.1]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 30 | 29 | 43 | 37
  Anti-PSW-135, Month 1 | 6.65 [4.29 to 10.3] | 0.15 [0.15 to 0.15] | 4.23 [2.94 to 6.09] | 8.17 [5.19 to 12.86]
  Anti-PSY, Month 1: number analyzed (Participants) | 30 | 27 | 43 | 37
  Anti-PSY, Month 1 | 10.37 [6.74 to 15.94] | 0.16 [0.15 to 0.17] | 8.07 [5.79 to 11.24] | 18.12 [12.41 to 26.46]
  Anti-PSA, Month 12: number analyzed (Participants) | 27 | 22 | 38 | 36
  Anti-PSA, Month 12 | 1.25 [0.68 to 2.3] | 0.17 [0.14 to 0.21] | 1.32 [0.9 to 1.95] | 4.43 [2.55 to 7.7]
  Anti-PSC, Month 12: number analyzed (Participants) | 27 | 27 | 39 | 37
  Anti-PSC, Month 12 | 0.39 [0.23 to 0.66] | 0.54 [0.34 to 0.86] | 0.28 [0.22 to 0.36] | 2.9 [1.94 to 4.35]
  Anti-PSW-135, Month 12: number analyzed (Participants) | 25 | 21 | 37 | 34
  Anti-PSW-135, Month 12 | 1.36 [1.06 to 1.74] | 0.21 [0.14 to 0.32] | 1.11 [0.79 to 1.57] | 3.16 [1.87 to 5.34]
  Anti-PSY, Month 12: number analyzed (Participants) | 26 | 21 | 37 | 35
  Anti-PSY, Month 12 | 2.36 [1.75 to 3.18] | 0.21 [0.14 to 0.33] | 1.84 [1.2 to 2.82] | 6.9 [4.51 to 10.54]

20. Secondary Outcome: Number of Seropositive and Seroprotected Subjects Against Different Meningococcal Serogroups
Description: A seropositive subject for rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY was defined as a vaccinated subject with antibody titers greater than or equal to (≥) 1:128, while for a seroprotected subject, titers were ≥1:8.
Time Frame: Before (PRE= at Month 12) and one month after (at Month 13) booster vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) Cohort for immune memory, which included subjects in the Toddlers subgroup from the ATP cohort for persistence, for whom assay results were available for antibodies against at least one study vaccine antigen component for the post-booster dose blood sampling.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 27 | 24
Participants
  rSBA-MenA ≥ 1:8, PRE: number analyzed (Participants) | 20 | 21
  rSBA-MenA ≥ 1:8, PRE | 20 | 17
  rSBA-MenC ≥ 1:8, PRE | 25 | 20
  rSBA-MenW-135 ≥ 1:8, PRE: number analyzed (Participants) | 27 | 23
  rSBA-MenW-135 ≥ 1:8, PRE | 26 | 9
  rSBA-MenY ≥ 1:8, PRE | 27 | 18
  rSBA-MenA ≥ 1:128, PRE: number analyzed (Participants) | 20 | 21
  rSBA-MenA ≥ 1:128, PRE | 20 | 16
  rSBA-MenC ≥ 1:128, PRE | 10 | 12
  rSBA-MenW-135 ≥ 1:128, PRE: number analyzed (Participants) | 27 | 23
  rSBA-MenW-135 ≥ 1:128, PRE | 23 | 4
  rSBA-MenY ≥ 1:128, PRE | 26 | 14
  rSBA-MenA ≥ 1:8, Month 13: number analyzed (Participants) | 6 | 20
  rSBA-MenA ≥ 1:8, Month 13 | 6 | 19
  rSBA-MenC ≥ 1:8, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenC ≥ 1:8, Month 13 | 25 | 24
  rSBA-MenW-135 ≥ 1:8, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenW-135 ≥ 1:8, Month 13 | 25 | 21
  rSBA-MenY ≥ 1:8, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenY ≥ 1:8, Month 13 | 25 | 22
  rSBA-MenA ≥ 1:128, Month 13: number analyzed (Participants) | 6 | 20
  rSBA-MenA ≥ 1:128, Month 13 | 6 | 19
  rSBA-MenC ≥ 1:128, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenC ≥ 1:128, Month 13 | 24 | 24
  rSBA-MenW-135 ≥ 1:128, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenW-135 ≥ 1:128, Month 13 | 25 | 18
  rSBA-MenY ≥ 1:128, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenY ≥ 1:128, Month 13 | 25 | 20

21. Secondary Outcome: Antibody Titers Against Different Meningococcal Serogroups
Description: as for outcome 4
Time Frame: Before (PRE= at Month 12) and one month after (at Month 13) booster vaccination
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 27 | 24
Titers
  rSBA-MenA, PRE: number analyzed (Participants) | 20 | 21
  rSBA-MenA, PRE | 2163.4 [1436.6 to 3257.9] | 175.7 [70.5 to 437.8]
  rSBA-MenC, PRE | 82.5 [50.3 to 135.4] | 102.5 [47.7 to 220.3]
  rSBA-MenW-135, PRE: number analyzed (Participants) | 27 | 23
  rSBA-MenW-135, PRE | 436 [243.7 to 780.2] | 15.5 [7 to 34.3]
  rSBA-MenY, PRE | 634.5 [420 to 958.3] | 93.6 [38.4 to 228.1]
  rSBA-MenA, Month 13: number analyzed (Participants) | 6 | 20
  rSBA-MenA, Month 13 | 3695.2 [1535.2 to 8894.7] | 984.6 [479.7 to 2021.2]
  rSBA-MenC, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenC, Month 13 | 7067.4 [4070.7 to 12270.3] | 9209.3 [5153.4 to 16457.5]
  rSBA-MenW-135, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenW-135, Month 13 | 5642.4 [3360 to 9475.4] | 255.6 [110.1 to 593.6]
  rSBA-MenY, Month 13: number analyzed (Participants) | 25 | 24
  rSBA-MenY, Month 13 | 3337.7 [2013.7 to 5532.1] | 323.8 [153.6 to 682.7]

22. Secondary Outcome: Number of Seropositive and Seroprotected Subjects Against Different Meningococcal Polysaccharides
Description: A seropositive subject for anti-PSA, anti-PSC, anti-PSW-135 and anti-PSY was defined as a vaccinated subject with antibody concentrations greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL), while for a seroprotected subject, antibody concentrations were ≥ 2.0 μg/mL.
Time Frame: Before (PRE= at Month 12) and one month after (at Month 13) booster vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 26 | 23
Participants
  Anti-PSA ≥ 0.3 μg/mL, PRE: number analyzed (Participants) | 24 | 19
  Anti-PSA ≥ 0.3 μg/mL, PRE | 19 | 1
  Anti-PSC ≥ 0.3 μg/mL, PRE: number analyzed (Participants) | 24 | 23
  Anti-PSC ≥ 0.3 μg/mL, PRE | 11 | 15
  Anti-PSW-135 ≥ 0.3 μg/mL, PRE: number analyzed (Participants) | 23 | 18
  Anti-PSW-135 ≥ 0.3 μg/mL, PRE | 23 | 2
  Anti-PSY ≥ 0.3 μg/mL, PRE: number analyzed (Participants) | 24 | 18
  Anti-PSY ≥ 0.3 μg/mL, PRE | 24 | 2
  Anti-PSA ≥ 2.0 μg/mL, PRE: number analyzed (Participants) | 24 | 19
  Anti-PSA ≥ 2.0 μg/mL, PRE | 7 | 0
  Anti-PSC ≥ 2.0 μg/mL, PRE: number analyzed (Participants) | 24 | 23
  Anti-PSC ≥ 2.0 μg/mL, PRE | 1 | 3
  Anti-PSW-135 ≥ 2.0 μg/mL, PRE: number analyzed (Participants) | 23 | 18
  Anti-PSW-135 ≥ 2.0 μg/mL, PRE | 5 | 1
  Anti-PSY ≥ 2.0 μg/mL, PRE: number analyzed (Participants) | 24 | 18
  Anti-PSY ≥ 2.0 μg/mL, PRE | 14 | 0
  Anti-PSA ≥ 0.3 μg/mL, Month 13: number analyzed (Participants) | 26 | 21
  Anti-PSA ≥ 0.3 μg/mL, Month 13 | 26 | 19
  Anti-PSC ≥ 0.3 μg/mL, Month 13: number analyzed (Participants) | 26 | 22
  Anti-PSC ≥ 0.3 μg/mL, Month 13 | 25 | 22
  Anti-PSW-135 ≥ 0.3 μg/mL, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSW-135 ≥ 0.3 μg/mL, Month 13 | 25 | 18
  Anti-PSY ≥ 0.3 μg/mL, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSY ≥ 0.3 μg/mL, Month 13 | 25 | 20
  Anti-PSA ≥ 2.0 μg/mL, Month 13: number analyzed (Participants) | 26 | 21
  Anti-PSA ≥ 2.0 μg/mL, Month 13 | 25 | 13
  Anti-PSC ≥ 2.0 μg/mL, Month 13: number analyzed (Participants) | 26 | 22
  Anti-PSC ≥ 2.0 μg/mL, Month 13 | 25 | 22
  Anti-PSW-135 ≥ 2.0 μg/mL, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSW-135 ≥ 2.0 μg/mL, Month 13 | 24 | 9
  Anti-PSY ≥ 2.0 μg/mL, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSY ≥ 2.0 μg/mL, Month 13 | 24 | 12

23. Secondary Outcome: Antibody Concentrations Against Different Meningococcal Polysaccharides
Description: as for outcome 7
Time Frame: Before (PRE= at Month 12) and one month after (at Month 13) booster vaccination
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 26 | 23
μg/mL
  Anti-PSA, PRE: number analyzed (Participants) | 24 | 19
  Anti-PSA, PRE | 0.98 [0.56 to 1.69] | 0.16 [0.14 to 0.18]
  Anti-PSC, PRE: number analyzed (Participants) | 24 | 23
  Anti-PSC, PRE | 1.33 [1.02 to 1.72] | 0.19 [0.13 to 0.27]
  Anti-PSW-135, PRE: number analyzed (Participants) | 23 | 18
  Anti-PSW-135, PRE | 25.67 [17.39 to 37.91] | 3.1 [1.34 to 7.2]
  Anti-PSY, PRE: number analyzed (Participants) | 24 | 18
  Anti-PSY, PRE | 56.94 [35.87 to 90.38] | 1.34 [0.63 to 2.88]
  Anti-PSA, Month 13: number analyzed (Participants) | 26 | 21
  Anti-PSA, Month 13 | 0.32 [0.22 to 0.48] | 0.5 [0.31 to 0.8]
  Anti-PSC, Month 13: number analyzed (Participants) | 26 | 22
  Anti-PSC, Month 13 | 2.34 [1.69 to 3.24] | 0.19 [0.13 to 0.26]
  Anti-PSW-135, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSW-135, Month 13 | 11.63 [7.73 to 17.5] | 15.23 [10.66 to 21.77]
  Anti-PSY, Month 13: number analyzed (Participants) | 25 | 21
  Anti-PSY, Month 13 | 79.03 [52.06 to 119.97] | 4.19 [2 to 8.78]

24. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 8-day (Days 0-7) post-vaccination period following booster dose
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all subjects who received the booster dose of Mencevax™ ACWY vaccine and had the symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 31 | 30
Participants
  Any Pain | 1 | 0
  Any Redness | 3 | 3
  Any Swelling | 1 | 1

25. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as rectal temperature equal to or above 38.0 degrees Celsius (°C)], irritability and loss of appetite. Any = incidence of a particular symptom regardless of intensity or relationship to vaccination.
Time Frame: During the 8-day (Days 0-7) post-vaccination period following booster dose
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 31 | 30
Participants
  Any Drowsiness | 3 | 5
  Any Fever (Rectally) | 5 | 3
  Any Irritability | 4 | 5
  Any Loss of appetite | 2 | 2

26. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) After the Primary Vaccination
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Days 0-30) after the primary meningococcal vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 54 | 50 | 52 | 52 | 52
Participants | 11 | 16 | 5 | 8 | 14 | 6 | 12 | 7 | 5 | 6

27. Secondary Outcome: Number of Subjects With Any Unsolicited AEs During the Primary Vaccination
Description: as for outcome 26
Time Frame: Within 31 days (Days 0-30) post-vaccination with diphteria, tetanus and acellular pertusis-containing vaccine, during the primary vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group
Number analyzed (Participants) | 38 | 40 | 37 | 40 | 39
Participants | 5 | 8 | 5 | 5 | 7

28. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: as for outcome 26
Time Frame: Within 31 days (Days 0-30) after the booster vaccination
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all subjects who received the booster dose of Mencevax™ ACWY vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group
Number analyzed (Participants) | 33 | 32
Participants | 3 | 5

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the primary vaccination study (from Month 0 up to Month 2)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group
Number analyzed (Participants) | 39 | 41 | 41 | 40 | 40 | 54 | 50 | 52 | 52 | 52
Participants | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 29
Time Frame: Since the last study contact in the primary study up to the end of the booster study (from Month 2 up to Month 13)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
Number analyzed (Participants) | 33 | 32 | 45 | 43
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 8-day (Days 0-7) post-vaccination period. Unsolicited AEs: within 31 days (Days 0-30) after each vaccination. SAEs: from the beginning of the primary study up to the end of the booster study (from Month 0 up to Month 13).
Description: The solicited local and general symptoms were only collected from those subjects who filled in their symptom sheets.
Arm/Group | GSK134612A Form1 (T), Primary Group | GSK134612A Form2 (T), Primary Group | GSK134612A Form3 (T), Primary Group | GSK134612A Form4 (T), Primary Group | Control (T), Primary Group | GSK134612A Form1 (C), Primary Group | GSK134612A Form2 (C), Primary Group | GSK134612A Form3 (C), Primary Group | GSK134612A Form4 (C), Primary Group | Control (C), Primary Group | GSK134612A Form1 (T), Booster Group | Control (T), Booster Group | GSK134612A Form1 (C), Booster Group | Control (C), Booster Group
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/41 | 0/40 | 0/40 | 0/54 | 0/50 | 0/52 | 0/52 | 0/52 | 0/33 | 0/32 | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/41 | 1/41 | 1/40 | 1/40 | 0/54 | 0/50 | 0/52 | 0/52 | 0/52 | 0/33 | 0/32 | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 20/39 | 27/41 | 23/41 | 24/40 | 25/40 | 10/54 | 11/50 | 10/52 | 11/52 | 13/52 | 5/33 | 5/32 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK134612A Form1 (T), Primary Group (N=39) | GSK134612A Form2 (T), Primary Group (N=41) | GSK134612A Form3 (T), Primary Group (N=41) | GSK134612A Form4 (T), Primary Group (N=40) | Control (T), Primary Group (N=40) | GSK134612A Form1 (C), Primary Group (N=54) | GSK134612A Form2 (C), Primary Group (N=50) | GSK134612A Form3 (C), Primary Group (N=52) | GSK134612A Form4 (C), Primary Group (N=52) | Control (C), Primary Group (N=52) | GSK134612A Form1 (T), Booster Group (N=33) | Control (T), Booster Group (N=32) | GSK134612A Form1 (C), Booster Group (N=45) | Control (C), Booster Group (N=43)
Maculo-papular rash (toddlers subgroup) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis (toddlers subgroup) (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (toddlers subgroup) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute bronchitis (toddlers subgroup) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK134612A Form1 (T), Primary Group (N=39) | GSK134612A Form2 (T), Primary Group (N=41) | GSK134612A Form3 (T), Primary Group (N=41) | GSK134612A Form4 (T), Primary Group (N=40) | Control (T), Primary Group (N=40) | GSK134612A Form1 (C), Primary Group (N=54) | GSK134612A Form2 (C), Primary Group (N=50) | GSK134612A Form3 (C), Primary Group (N=52) | GSK134612A Form4 (C), Primary Group (N=52) | Control (C), Primary Group (N=52) | GSK134612A Form1 (T), Booster Group (N=33) | Control (T), Booster Group (N=32) | GSK134612A Form1 (C), Booster Group (N=0) | Control (C), Booster Group (N=0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 2 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1 | 0/0 | 0/0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0/0 | 0/0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pain (GSK134612A conjugate vaccine) (General disorders) | 4/38 | 8 | 3/39 | 6 | 4/39 | 10/52 | 11 | 9/50 | 11 | 13/51 | 1/31 | 0/30 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Pain (Infanrix™-containing vaccine) (General disorders) | 3/38 | 10/39 | 6/37 | 7/39 | 6/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (GSK134612A conjugate vaccine) (General disorders) | 9/38 | 12 | 10/39 | 9 | 11/39 | 9/52 | 11 | 10/50 | 9 | 7/51 | 3/31 | 3/30 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Redness (Infanrix™-containing vaccine) (General disorders) | 7/38 | 13/39 | 9/37 | 8/39 | 7/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (GSK134612A conjugate vaccine) (General disorders) | 1/38 | 6 | 7/39 | 6 | 4/39 | 7/52 | 9 | 8/50 | 10 | 4/51 | 1/31 | 1/30 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Swelling (Infanrix™-containing vaccine) (General disorders) | 3/38 | 7/39 | 9/37 | 7/39 | 3/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited local symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (GSK134612A conjugate vaccine) (General disorders) | 1/38 | 5 | 4/39 | 4 | 5/39 | 4/52 | 2 | 0/50 | 5 | 4/51 | 3/31 | 5/30 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Drowsiness (Infanrix™-containing vaccine) (General disorders) | 2/38 | 2/39 | 3/37 | 7/39 | 3/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Axillary/Rectally fever (GSK134612A conjugate vaccine) (General disorders) | 5/38 | 8 | 8/39 | 3 | 5/39 | 4/52 | 4 | 3/50 | 3 | 3/51 | 5/31 | 3/30 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Axillary fever (Infanrix™-containing vaccine) (General disorders) | 4/38 | 5/39 | 5/37 | 5/39 | 8/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (GSK134612A conjugate vaccine) (General disorders) | 4/38 | 9 | 6/39 | 5 | 5/39 | 2/52 | 4 | 2/50 | 4 | 7/51 | 4/31 | 5/30 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Irritability (Infanrix™-containing vaccine) (General disorders) | 6/38 | 7/39 | 3/37 | 9/39 | 5/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (GSK134612A conjugate vaccine) (General disorders) | 1/38 | 6 | 5/39 | 3 | 6/39 | 2/52 | 3 | 2/50 | 6 | 3/51 | 2/31 | 2/30 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.
Loss of appetite (Infanrix™-containing vaccine) (General disorders) | 4/38 | 3/39 | 2/37 | 6/39 | 2/37 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 — This solicited general symptom was only collected from subjects with their symptom sheets completed.

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.